CLINICAL TRIAL: NCT06330337
Title: Specific Model Electroacupuncture Stimulation Promotes Paclitaxel Delivery Across the BBB for Postoperative Glioma Patients: A Randomized Controlled Study
Brief Title: Effect of Electroacupuncture Combined With Paclitaxel Clinical Efficacy of Patients With Recurrence of High-grade Glioma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xianming Lin, Clinical Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZSLL-KY-2024-010-01
Record Dates: First submitted 2024-02-26; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Glioma
Keywords: glioma; Specific Mode Electroacupuncture Stimulation; protein-bound paclitaxel; blood-brain barrier
MeSH Terms: conditions — Glioma | interventions — Administration, Oral; Infusions, Intravenous; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMZ group (Other): Temozolomide（TMZ） was given orally or intravenously 150mg/(m2·d) for 5 days, repeated every 28 days for 6 cycles
  Interventions: Drug: Temozolomide（TMZ） injection or oral administration
- SMES+ABX+TMZ Group (Other): Drug:
  Oral or intravenous infusion of TMZ 150mg/(m2·d) for 5 days, repeated after 23 days of suspension, a total of 6 treatment cycles. During the TMZ treatment cycle, specific mode electroacupuncture stimulation（SMES） combined with Paclitaxel for Injection (Albumin Bound)（ABX） were used on day 1 and day 8.
  ABX： ABX was prepared with 0.9% sodium chloride injection and the dosage required by the patient was calculated at 110mg/mm2. Then the intravenous infusion continues for 30 minutes.
  SMES：Immediately after the ABX intravenous infusion began, the patient was placed in a supine position, the skin was routinely disinfected with 75% ethanol, and a stainless steel needle was inserted into GV20 and GV26.Then, the needles are stimulated by using an acupuncture point nerve stimulator with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off).
  Interventions: Drug: Temozolomide（TMZ） injection or oral administration; Drug: Albumin-Bound Paclitaxel(ABX) intravenous drip; Device: Specific mode electroacupuncture stimulation(SMES) intervention

INTERVENTIONS:
Drug: Temozolomide（TMZ） injection or oral administration — Oral administration of TMZ150-200mg/m2/ day, continuous use for 5 days, discontinued for 23 days, for a treatment cycle, a total of 6 cycles.
Drug: Albumin-Bound Paclitaxel(ABX) intravenous drip — ABX was administered intravenously at a dose of 110mg/m2 on days 1 and 8 of a 28-day treatment cycle
  Arms: SMES+ABX+TMZ Group
Device: Specific mode electroacupuncture stimulation(SMES) intervention — Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle (size 0.25mm×40mm, Hua Tuo brand, Suzhou Medical Supplies Company Ltd in Jiangsu, China) will be inserted in GV20（Baihui) and the stainless needle(size 0.25mm×25mm, described above) will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness (the reaction of "De Qi"). Then, the needles are stimulated by using an acupuncture point nerve stimulator (HANS-200, Nanjing Jinsheng, Ltd., China) with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off).The 28-day treatment cycle was followed by simultaneous intervention with ABX on days 1 and 8.
  Arms: SMES+ABX+TMZ Group

SUMMARY:
Gliomas are the most common type of primary brain tumors, with surgery followed by radiotherapy and chemotherapy as the main treatment modalities. However, they are highly prone to recurrence, presenting significant treatment challenges, especially for high-grade gliomas, which have a 5-year survival rate of only 5.5%. Paclitaxel, a common chemotherapeutic agent, exhibits antitumor effects in vitro that are 1400 times stronger than those of temozolomide (the first-line chemotherapy drug for gliomas). However, due to its large molecular weight (approximately 893 Da), it cannot cross the blood-brain barrier, precluding its use as a first-line treatment for gliomas. Preliminary research by our team has demonstrated that Specific Mode Electroacupuncture Stimulation (SMES) can open the blood-brain barrier, enhancing the concentration of albumin-bound paclitaxel (ABX) in tumor tissues, peritumoral tissues, and surrounding invasive tissues, thereby exerting antitumor effects. Consequently, this study aims to observe the safety and efficacy of SMES combined with ABX in treating patients with recurrent high-grade gliomas postoperatively, to explore its mechanisms of action, extend survival, improve quality of life, and forge new theories and methods for the integrative treatment of brain tumors combining traditional Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed high-grade glioma, with standard radiotherapy and chemotherapy post-surgical resection deemed unsuccessful, and recurrence confirmed by imaging.
2. Age ≥18 and ≤70 years, open to all genders.
3. If receiving dexamethasone for mass effect, a stable daily dose of <6 mg in the 7 days prior to enrollment, or if the dose of dexamethasone is decreasing, an average daily dose of <6 mg in the 7 days prior to enrollment. Patients receiving dexamethasone for reasons other than mass effect are still eligible.
4. A Karnofsky Performance Score (KPS) ≥70 or a World Health Organization (WHO) performance status of ≤2.
5. Meets the criteria for acupuncture, with no severe complications, able to undergo acupuncture treatment and demonstrates good compliance.
6. Clear consciousness, with the ability to perceive and distinguish pain, and capable of basic communication.
7. Signed informed consent, voluntarily participating in this study.

Exclusion Criteria:

1. Uncontrolled epileptic seizures;
2. Peripheral neuropathy > Grade 1;
3. Currently participating in another clinical trial or having participated in a clinical trial that concluded less than 3 months ago;
4. Previous treatment with paclitaxel or similar chemotherapeutic or biologic agents, or history of allergic reactions to these compounds;
5. Patients with severe cardiac, hepatic, renal, or hematologic dysfunction (criteria within 14 days prior to treatment include: a. Hemoglobin ≥ 90.0 g/L; b. White blood cells ≥ 3.010^9/L; c. Absolute neutrophil count ≥ 1500/µL; d. Platelets ≥ 10010^9/µL; e. Total bilirubin (TbIL) ≤5.0 x ULN; f. Serum aspartate aminotransferase (SGOT) ≤10 x ULN and TbIL >3 to ≤5.0 x ULN; g. Creatinine ≤1.5 mg/dL, estimated creatinine clearance ≥ 30 mL/min to <90 mL/min);
6. Pregnant or breastfeeding women;
7. Individuals with cognitive impairments such as congenital dementia, or with histories of alcohol, drug, or psychotropic substance abuse;
8. Individuals with a history of needle fainting or infections at the site of acupuncture;
9. Patients with conductive foreign bodies within the body;
10. Individuals unable to undergo enhanced MRI examinations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival（OS） | Starting from randomization, during the follow-up phase, telephone follow-ups to record survival status are conducted every two months, totaling six follow-ups. This structured approach ensures a comprehensive assessment of patient out
  The duration from randomization to death due to any cause is measured (for patients lost to follow-up, the last follow-up date is used; for patients alive at the end of the study, the date of the last follow-up is considered).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 12 months were assessed from the date of randomization to the date of first recording to the date of progression or the date of death from any cause, whichever came first
  The period from randomization to the first occurrence of tumor progression or death is meticulously monitored.
Head MRI (plain and enhanced) | One treatment cycle is 28 days, with cranial MRI scans conducted one day before the start of treatment cycles 1, 3, and 5, and at the end of treatment cycle 6.
  The short-term efficacy of the two groups is analyzed, referencing the RANO criteria for assessing the efficacy of solid tumor treatment before and after therapy. Complete Response (CR) is when visible tumor lesions disappear completely, maintained for >4 weeks (in accordance with RANO criteria and RECIST version 2000). Partial Response (PR) involves a reduction of ≥50% in the sum of the diameters of the tumor lesions, with no increase in other lesions and no new lesions appearing, maintained for >4 weeks. Stable Disease (SD) is defined as the sum of the diameters of the tumor lesions decreasing by <50% or increasing by ≤25%, with no new lesions appearing, maintained for >4 weeks. Progression (PD) occurs when there is an increase of >25% in the sum
he Karnofsky Performance Score (KPS) | One treatment cycle is 28 days, with assessments conducted one day before the start of treatment cycles 1 through 6 and one day before the end of treatment cycle 6.
  KPS ranges from 0 to 100, with scores directly correlating to quality of life.
The Eastern Cooperative Oncology Group (ECOG) | One treatment cycle is 28 days, with assessments conducted one day before the start of treatment cycles 1 through 6 and one day before the end of treatment cycle 6.
  ECOG Performance Status is scored from 0 to 5, with scores inversely related to quality of life.
The Quality of Life (QOL) | One treatment cycle is 28 days, with assessments conducted one day before the start of treatment cycles 1 through 6 and one day before the end of treatment cycle 6.
  QOL scale for cancer patients assesses quality of life, with a total score ranging from 0 to 60, where scores directly correlate with quality of life.
The Neurological Assessment for Neuro-Oncology (NANO) | One treatment cycle is 28 days, with assessments conducted one day before the start of treatment cycles 1 through 6 and one day before the end of treatment cycle 6.
  NANO Scale quantitatively assesses nine neurological functions in patients, including gait, muscle strength, sensation, visual fields, facial strength, speech, cognition, and limb coordination, with each category scored between 0 to 3 or 0 to 2.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data and results of this study need to be confirmed by Lin Xianming

REFERENCES:
- [Result] Weller M, Wick W, Aldape K, Brada M, Berger M, Pfister SM, Nishikawa R, Rosenthal M, Wen PY, Stupp R, Reifenberger G. Glioma. Nat Rev Dis Primers. 2015 Jul 16;1:15017. doi: 10.1038/nrdp.2015.17. PMID 27188790
- [Result] Rapp M, Baernreuther J, Turowski B, Steiger HJ, Sabel M, Kamp MA. Recurrence Pattern Analysis of Primary Glioblastoma. World Neurosurg. 2017 Jul;103:733-740. doi: 10.1016/j.wneu.2017.04.053. Epub 2017 Apr 19. PMID 28434963
- [Result] Wick W, Stupp R, Beule AC, Bromberg J, Wick A, Ernemann U, Platten M, Marosi C, Mason WP, van den Bent M, Weller M, Rorden C, Karnath HO; European Organisation for Research and Treatment of Cancer and the National Cancer Institute of Canada Clinical Trials Group. A novel tool to analyze MRI recurrence patterns in glioblastoma. Neuro Oncol. 2008 Dec;10(6):1019-24. doi: 10.1215/15228517-2008-058. Epub 2008 Jul 31. PMID 18676355
- [Result] Stupp R, Hegi ME, Mason WP, van den Bent MJ, Taphoorn MJ, Janzer RC, Ludwin SK, Allgeier A, Fisher B, Belanger K, Hau P, Brandes AA, Gijtenbeek J, Marosi C, Vecht CJ, Mokhtari K, Wesseling P, Villa S, Eisenhauer E, Gorlia T, Weller M, Lacombe D, Cairncross JG, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumour and Radiation Oncology Groups; National Cancer Institute of Canada Clinical Trials Group. Effects of radiotherapy with concomitant and adjuvant temozolomide versus radiotherapy alone on survival in glioblastoma in a randomised phase III study: 5-year analysis of the EORTC-NCIC trial. Lancet Oncol. 2009 May;10(5):459-66. doi: 10.1016/S1470-2045(09)70025-7. Epub 2009 Mar 9. PMID 19269895
- [Result] Dmello C, Sonabend A, Arrieta VA, Zhang DY, Kanojia D, Chen L, Gould A, Zhang J, Kang SJ, Winter J, Horbinski C, Amidei C, Gyorffy B, Cordero A, Chang CL, Castro B, Hsu P, Ahmed AU, Lesniak MS, Stupp R, Sonabend AM. Translocon-associated Protein Subunit SSR3 Determines and Predicts Susceptibility to Paclitaxel in Breast Cancer and Glioblastoma. Clin Cancer Res. 2022 Jul 15;28(14):3156-3169. doi: 10.1158/1078-0432.CCR-21-2563. PMID 35552677
- [Result] Aldape K, Brindle KM, Chesler L, Chopra R, Gajjar A, Gilbert MR, Gottardo N, Gutmann DH, Hargrave D, Holland EC, Jones DTW, Joyce JA, Kearns P, Kieran MW, Mellinghoff IK, Merchant M, Pfister SM, Pollard SM, Ramaswamy V, Rich JN, Robinson GW, Rowitch DH, Sampson JH, Taylor MD, Workman P, Gilbertson RJ. Challenges to curing primary brain tumours. Nat Rev Clin Oncol. 2019 Aug;16(8):509-520. doi: 10.1038/s41571-019-0177-5. PMID 30733593
- [Result] Terstappen GC, Meyer AH, Bell RD, Zhang W. Strategies for delivering therapeutics across the blood-brain barrier. Nat Rev Drug Discov. 2021 May;20(5):362-383. doi: 10.1038/s41573-021-00139-y. Epub 2021 Mar 1. PMID 33649582
- [Result] Parrish KE, Sarkaria JN, Elmquist WF. Improving drug delivery to primary and metastatic brain tumors: strategies to overcome the blood-brain barrier. Clin Pharmacol Ther. 2015 Apr;97(4):336-46. doi: 10.1002/cpt.71. Epub 2015 Feb 18. PMID 25669487
- [Result] Cardoso FL, Brites D, Brito MA. Looking at the blood-brain barrier: molecular anatomy and possible investigation approaches. Brain Res Rev. 2010 Sep 24;64(2):328-63. doi: 10.1016/j.brainresrev.2010.05.003. Epub 2010 May 26. PMID 20685221
- [Result] Agarwal S, Sane R, Oberoi R, Ohlfest JR, Elmquist WF. Delivery of molecularly targeted therapy to malignant glioma, a disease of the whole brain. Expert Rev Mol Med. 2011 May 13;13:e17. doi: 10.1017/S1462399411001888. PMID 21676290
- [Result] Fowler MJ, Cotter JD, Knight BE, Sevick-Muraca EM, Sandberg DI, Sirianni RW. Intrathecal drug delivery in the era of nanomedicine. Adv Drug Deliv Rev. 2020;165-166:77-95. doi: 10.1016/j.addr.2020.02.006. Epub 2020 Mar 3. PMID 32142739
- [Result] Malani R, Fleisher M, Kumthekar P, Lin X, Omuro A, Groves MD, Lin NU, Melisko M, Lassman AB, Jeyapalan S, Seidman A, Skakodub A, Boire A, DeAngelis LM, Rosenblum M, Raizer J, Pentsova E. Cerebrospinal fluid circulating tumor cells as a quantifiable measurement of leptomeningeal metastases in patients with HER2 positive cancer. J Neurooncol. 2020 Jul;148(3):599-606. doi: 10.1007/s11060-020-03555-z. Epub 2020 Jun 6. PMID 32506369
- [Result] Zagouri F, Zoumpourlis P, Le Rhun E, Bartsch R, Zografos E, Apostolidou K, Dimopoulos MA, Preusser M. Intrathecal administration of anti-HER2 treatment for the treatment of meningeal carcinomatosis in breast cancer: A metanalysis with meta-regression. Cancer Treat Rev. 2020 Aug;88:102046. doi: 10.1016/j.ctrv.2020.102046. Epub 2020 Jun 3. PMID 32599393
- [Result] Tosi U, Kommidi H, Adeuyan O, Guo H, Maachani UB, Chen N, Su T, Zhang G, Pisapia DJ, Dahmane N, Ting R, Souweidane MM. PET, image-guided HDAC inhibition of pediatric diffuse midline glioma improves survival in murine models. Sci Adv. 2020 Jul 24;6(30):eabb4105. doi: 10.1126/sciadv.abb4105. eCollection 2020 Jul. PMID 32832670
- [Result] Graham-Gurysh EG, Murthy AB, Moore KM, Hingtgen SD, Bachelder EM, Ainslie KM. Synergistic drug combinations for a precision medicine approach to interstitial glioblastoma therapy. J Control Release. 2020 Jul 10;323:282-292. doi: 10.1016/j.jconrel.2020.04.028. Epub 2020 Apr 23. PMID 32335153
- [Result] Siegal T, Rubinstein R, Bokstein F, Schwartz A, Lossos A, Shalom E, Chisin R, Gomori JM. In vivo assessment of the window of barrier opening after osmotic blood-brain barrier disruption in humans. J Neurosurg. 2000 Apr;92(4):599-605. doi: 10.3171/jns.2000.92.4.0599. PMID 10761648
- [Result] Park J, Aryal M, Vykhodtseva N, Zhang YZ, McDannold N. Evaluation of permeability, doxorubicin delivery, and drug retention in a rat brain tumor model after ultrasound-induced blood-tumor barrier disruption. J Control Release. 2017 Mar 28;250:77-85. doi: 10.1016/j.jconrel.2016.10.011. Epub 2016 Oct 11. PMID 27742444
- [Result] Chen Zhongjian, Zhang Yuan, Zheng Yejiao, Yang Haiyan, Gu Liqiang. Research Progress on Borneol Promoting Drug Permeation Through the Blood-Brain Barrier [J]. Chinese Traditional Patent Medicine, 2019, 41(09): 2170-2173.
- [Result] Guo Junqia, Zhang Rong, Duan Meimei, Xing Yanmei. The Effect of Natural Borneol on the Permeability of MTX Through the Blood-Tumor Barrier [J]. Traditional Chinese Drug Research & Clinical Pharmacology, 2015, 26(01): 73-77.
- [Result] Zhang S, Gong P, Zhang J, Mao X, Zhao Y, Wang H, Gan L, Lin X. Specific Frequency Electroacupuncture Stimulation Transiently Enhances the Permeability of the Blood-Brain Barrier and Induces Tight Junction Changes. Front Neurosci. 2020 Oct 6;14:582324. doi: 10.3389/fnins.2020.582324. eCollection 2020. PMID 33122995
- [Result] Caffery B, Lee JS, Alexander-Bryant AA. Vectors for Glioblastoma Gene Therapy: Viral & Non-Viral Delivery Strategies. Nanomaterials (Basel). 2019 Jan 16;9(1):105. doi: 10.3390/nano9010105. PMID 30654536
- [Result] Barretina J, Caponigro G, Stransky N, Venkatesan K, Margolin AA, Kim S, Wilson CJ, Lehar J, Kryukov GV, Sonkin D, Reddy A, Liu M, Murray L, Berger MF, Monahan JE, Morais P, Meltzer J, Korejwa A, Jane-Valbuena J, Mapa FA, Thibault J, Bric-Furlong E, Raman P, Shipway A, Engels IH, Cheng J, Yu GK, Yu J, Aspesi P Jr, de Silva M, Jagtap K, Jones MD, Wang L, Hatton C, Palescandolo E, Gupta S, Mahan S, Sougnez C, Onofrio RC, Liefeld T, MacConaill L, Winckler W, Reich M, Li N, Mesirov JP, Gabriel SB, Getz G, Ardlie K, Chan V, Myer VE, Weber BL, Porter J, Warmuth M, Finan P, Harris JL, Meyerson M, Golub TR, Morrissey MP, Sellers WR, Schlegel R, Garraway LA. The Cancer Cell Line Encyclopedia enables predictive modelling of anticancer drug sensitivity. Nature. 2012 Mar 28;483(7391):603-7. doi: 10.1038/nature11003. PMID 22460905
- [Result] Chang SM, Kuhn JG, Robins HI, Schold SC Jr, Spence AM, Berger MS, Mehta M, Pollack IF, Rankin C, Prados MD. A Phase II study of paclitaxel in patients with recurrent malignant glioma using different doses depending upon the concomitant use of anticonvulsants: a North American Brain Tumor Consortium report. Cancer. 2001 Jan 15;91(2):417-22. doi: 10.1002/1097-0142(20010115)91:23.0.co;2-9. PMID 11180089
- [Result] Chamberlain MC, Kormanik P. Salvage chemotherapy with paclitaxel for recurrent primary brain tumors. J Clin Oncol. 1995 Aug;13(8):2066-71. doi: 10.1200/JCO.1995.13.8.2066. PMID 7636549
- [Result] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Result] Sonabend AM, Gould A, Amidei C, Ward R, Schmidt KA, Zhang DY, Gomez C, Bebawy JF, Liu BP, Bouchoux G, Desseaux C, Helenowski IB, Lukas RV, Dixit K, Kumthekar P, Arrieta VA, Lesniak MS, Carpentier A, Zhang H, Muzzio M, Canney M, Stupp R. Repeated blood-brain barrier opening with an implantable ultrasound device for delivery of albumin-bound paclitaxel in patients with recurrent glioblastoma: a phase 1 trial. Lancet Oncol. 2023 May;24(5):509-522. doi: 10.1016/S1470-2045(23)00112-2. PMID 37142373